CLINICAL TRIAL: NCT04005690
Title: A Window of Opportunity Strategy for Targeted Pathway Inhibition in Patients With Pancreatic Ductal Adenocarcinoma
Brief Title: Targeted Pathway Inhibition in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: American Association for Cancer Research (Other); Oregon Health and Science University (Other); Genentech, Inc. (Industry); Cardiff Oncology (Industry)
Responsible Party: Principal Investigator, Charles D Lopez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019211; NCI-2019-01265 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019211 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-05-23; First posted 2019-07-02 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Ductal Adenocarcinoma; Borderline Resectable Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — cobimetinib; olaparib; onvansertib; AZD5305; tremelimumab; Immunoglobulin G; Antigens; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm Olaparib (Experimental): Patients receive olaparib PO BID on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)
  Interventions: Drug: Olaparib
- Arm Cobimetinib (Experimental): Patients receive cobimetinib PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)
  Interventions: Drug: Cobimetinib
- Arm Onvansertib (Experimental): Patients receive onvansertib PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)
  Interventions: Drug: Onvansertib
- Arm Azenosertib (Experimental): Patients receive azenosertib PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.
  Interventions: Drug: Azenosertib
- Arm AZD5305 (Experimental): Patients receive AZD5305 PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.
  Interventions: Drug: Saruparib
- Arm Tremelimumab (Experimental): Patients receive tremelimumab IV over 60 minutes one-time. Within 12-24 hours of cycle completion, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.
  Interventions: Biological: Tremelimumab

INTERVENTIONS:
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
  Arms: Arm Cobimetinib
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
  Arms: Arm Olaparib
Drug: Onvansertib — Given PO
  Other Names: 'PLK1 Inhibitor PCM-075; NMS-1286937; PCM 075; PCM-075; PLK-1 Inhibitor PCM-075; Polo-like Kinase 1 Inhibitor NMS-1286937; Polo-like Kinase 1 Inhibitor PCM-075
  Arms: Arm Onvansertib
Drug: Azenosertib — Given PO
  Other Names: ZN-c3; KP-2638; C29H34N8O2
  Arms: Arm Azenosertib
Drug: Saruparib — Given PO
  Other Names: AZD5305; 2589531-76-8; AZD 5305; AZD-5305; PARP Inhibitor AZD5305
  Arms: Arm AZD5305
Biological: Tremelimumab — Given IV
  Other Names: 745013-59-6; Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP 675; CP 675206; CP-675; CP-675,206; CP-675206; CP675; CP675206; Imjudo; Immunoglobulin G2; Anti-(Human CTLA-4 (Antigen)) (Human Monoclonal CP-675206 Clone 11.2.1 Heavy Chain) Disulfide with Human Monoclonal CP-675206 Clone 11.2.1 Light Chain; Dimer; ticilimumab; Tremelimumab-actl
  Arms: Arm Tremelimumab

SUMMARY:
This early phase I trial aims to determine how cobimetinib, olaparib, onvansertib, azenosertib, AZD5305 or tremelimumab works in patients with pancreatic cancer. Validation of cobimetinib, olaparib, onvansertib azenosertib, AZD5305 and tremelimumab molecular targets will be explored by comparing pre-treatment biopsies with post-treatment specimens. This knowledge will help design future biomarker driven trials to determine whether giving cobimetinib, or olaparib, or onvansertib or azenosertib, or AZD5305, or tremelimumab will work better than standard treatments in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Independently assess the pharmacodynamic (PD) feasibility of detecting a measurable change in tumor biology at post-treatment from baseline (i.e., before the study treatment window) for all feasibility-evaluable participants in each study arm.

SECONDARY OBJECTIVE:

I. Assess preliminary safety and tolerability of the proposed study agent(s) in each study arm.

EXPLORATORY OBJECTIVES:

I. Identify predictive biomarkers of sensitivity to assigned study agent(s).

II. Identify emerging mechanism(s) of resistance to assigned study agent(s).

III. Determine cellular and molecular changes in pancreatic tumor cells exposed to assigned study agent(s).

IV. Identify tumor markers suggestive of combinatorial therapy that could overcome resistance to therapy.

OUTLINE: Patients are assigned to 1 of 6 arms.

ARM Olaparib: Patients receive olaparib orally (PO) twice daily (BID) on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)

ARM Cobimetinib: Patients receive cobimetinib PO once daily (QD) on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)

ARM Onvansertib: Patients receive onvansertib PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease. (Arm Closed as of 8/12/2024)

ARM Azenosertib: Patients receive azenosertib PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.

ARM AZD5305: Patients receive AZD5305 (saruparib) PO QD on days 1-10 in the absence of disease progression or unacceptable toxicity. Within 12-24 hours, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.

ARM Tremelimumab: Patients receive tremelimumab intravenously (IV) over 60 minutes one-time. Within 12-24 hours of cycle completion, patients undergo biopsy or surgery as clinically appropriate per institutional standards for management of patient's disease.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Clinically-confirmed diagnosis of resectable, borderline resectable, locally-advanced or metastatic adenocarcinoma of the pancreas.

  * Patients with disease that is eligible for curative surgery may not be eligible for all study arms.
  * Participants may be treatment naïve or have received prior therapy for the treatment of their pancreatic ductal adenocarcinoma (PDAC). A minimum washout period of 10-days after completing the most recent line of therapy is required before a participant can initiate treatment with study agent(s)
* Based on available imaging, participant must have at least one disease lesion that can be biopsied in accordance with institutional standards
* Hemoglobin >= 9.0 g/dL with no blood transfusion within 28 days of starting treatment (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion
* White blood cells (WBC) > 3 x 10^9/L (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3) (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion.

  * May be waived on a case-by-case basis for patient populations recognized to have normal baseline values below this level
* Platelet count >= 100 x 10^9/L (> 100,000 per mm^3) (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion
* Creatinine =< 1.5 x upper limit of normal (ULN), OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min/1.73m^2 for participants with creatinine levels > 1.5 x institutional ULN (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion.

  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (within 4 weeks prior to initiating window treatment). Note: laboratory tests performed after initial screening (but still within the screening window) will be evaluated by the investigator; should any of these values fall outside eligibility parameters, the patient may still be eligible per investigator discretion
* Participants must be willing to undergo mandatory on-study tumor biopsies
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Participant must be able to swallow tablets or capsules. A participant with any gastrointestinal disease that would impair ability to swallow, retain, or absorb drug is not eligible
* Participants of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants must agree to use an adequate method of contraception starting with the first dose of study therapy and for the required length of time ascribed to the assigned study drug assignment
* No other prior invasive malignancy is allowed except for the following: adequately treated basal (or squamous cell) skin cancer, in situ breast or cervical cancer, any malignancy treated with a curative intent without evidence of disease recurrence for at least 6 months
* Individuals must not have known active hepatitis B virus (HBV). Those who have completed curative therapy for hepatitis C virus (HCV) are eligible. HCV infection permitted but patient must be Child's Pugh A. Patients with known human immunodeficiency virus (HIV) infection are eligible if they meet all of the following 3 criteria:

  * CD4 counts >= 350 mm^3
  * Serum HIV viral load of < 25,000 IU/ml and
  * Treated on a stable antiretroviral regimen
  * Note: HIV testing is not required at screening, unless if required by local regulations, where the testing will be done by local laboratory
* AZENOSERTIB SPECIFIC CRITERIA: Those with prior treatment with a WEE1 inhibitor are not eligible
* AZENOSERTIB SPECIFIC CRITERIA: Patients are not eligible if any of the following treatment interventions have occurred within the specified time frame(s) prior to starting study intervention:

  * Major surgery within 28 days (the surgical incision should be fully healed prior to study drug administration)
  * Radiation therapy within 21 days; however, if the radiation portal covered ≤ 5% of the bone marrow reserve, the subject is eligible irrespective of the end date of radiotherapy
  * Autologous or allogeneic stem cell transplant within 3 months
  * Current use of an investigational agent that is not expected to be cleared by the first dosing of study drug or that has demonstrated to have prolonged side effects
  * Prescription, non-prescription drugs or food known as moderate to strong inducers of CYP3A within 2 weeks
* AZENOSERTIB SPECIFIC CRITERIA: Patients are not eligible if there is a serious illness or medical condition(s) including, but not limited to, the following:

  * Symptomatic brain metastases
  * Leptomeningeal disease that requires or is anticipated to require immediate treatment.
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the subject inappropriate for entry into this study
  * Significant gastrointestinal abnormalities, including an inability to take oral medication, requirement for IV alimentation, active peptic ulcer, chronic diarrhea or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption
  * Active or uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥ 72 hours
* AZENOSERTIB SPECIFIC CRITERIA: 12-lead ECG demonstrating a corrected QT interval using Fridericia's formula (QTcF) of >480 ms, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid
* AZENOSERTIB SPECIFIC CRITERIA: History or current evidence of congenital or family history of long QT syndrome or Torsade de Pointes
* AZENOSERTIB SPECIFIC CRITERIA: Patients are not eligible in cases of unresolved toxicity of grade > 1 attributed to any prior therapies (excluding grade 2 neuropathy, alopecia or skin pigmentation)
* AZENOSERTIB SPECIFIC CRITERIA: Patients are not eligible if there is known hypersensitivity to any drugs similar to ZN-c3 in class
* AZENOSERTIB SPECIFIC CRITERIA: Individuals that are pregnant or breast-feeding are not eligible
* AZENOSERTIB SPECIFIC CRITERIA: Participants must agree to use an adequate method of contraception as follows:

  * Participants of childbearing potential agree to use adequate methods of contraception for the duration of study participation.
  * Sperm-producing participants must agree to refrain from sperm donation during the study and for 30 days after the last dose of study drug
* AZENOSERTIB SPECIFIC CRITERIA: Participant requiring any medications that can lead to significant QT prolongation are not eligible
* AZENOSERTIB SPECIFIC CRITERIA: Participant requires administration of strong and moderate CYP3A4 inhibitors and inducers as well as strong and moderate P-glycoprotein (P-gp) inhibitors are not eligible
* AZENOSERTIB SPECIFIC CRITERIA: Due to potential CYP3A4 interaction with the study medication, participants are asked to refrain from consumption of seville oranges, grapefruit or grapefruit juice, ppomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices) from 7 days prior to the initiating study agent and during the entire study. NOTE: Orange juice is permitted
* AZD5305 SPECIFIC CRITERIA: Participants must agree to use an adequate method of contraception as follows:

  * Participants of childbearing potential must agree to use adequate methods of contraception starting with the first dose of study therapy through at least 6 months after the last dose of study therapy
  * Sperm-producing participants must use a condom during treatment and for 6 months after the last dose of AZD5305 when having sexual intercourse with an individual that is pregnant or of childbearing potential. Individuals that are partners of sperm-producing participants should also use a highly effective form of contraception if they are of childbearing potential
* TREMELIMUMAB SPECIFIC CRITERIA: Participants of childbearing potential must agree to use adequate methods of contraception starting with the first dose of study therapy through at least 3 months after the last dose of study therapy

Exclusion Criteria:

* Tumor not accessible for core biopsy
* Medical co-morbidities that are deemed to make risk of surgery unacceptably high as determined by institutional standards
* Recent major surgery within 4 weeks prior to starting study treatment. Minor surgery within 2 weeks of starting study treatment. Patients must be recovered from effects of surgery
* Concomitant use of known strong (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, modafinil)
* Concomitant use of known strong CYP3A inhibitors (e.g., itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g., ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil)
* Concomitant use of other anti-cancer therapy (chemotherapy, immunotherapy, hormonal therapy (hormone replacement therapy is acceptable), radiotherapy (except for palliative), biological therapy or other novel agent) or live virus and live bacterial vaccines while the patient is receiving study medication. Strong or moderate CYP3A inhibitors and inducers should not be taken with study treatment; however, if no other suitable alternative concomitant medication is available, dose reductions may be allowed under careful monitoring
* Known severe hypersensitivity to the study agent(s) (or equivalent agents, respectively), or any excipient of these medicinal products, or history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agent(s)
* Clinically significant cardiac disease or impaired cardiac function, including any of the following:

  * Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade >= 2) uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment
  * Corrected QT using Fridericia's formula (QTcF) > 470 msec for females, or > 450 msec for males, on screening electrocardiogram (ECG) or congenital long QT syndrome
  * Acute myocardial infarction or unstable angina pectoris < 6 months prior to screening
* Clinically significant cardiac disease or impaired cardiac function
* Female participant who is pregnant or lactating
* Participant is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Participant has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Psychiatric illness/social situations that would limit compliance with study requirements
* Participants with a history of hypersensitivity reactions to study agents or their excipients
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through at least 120 days after the last dose of trial treatment
* AZD5305 SPECIFIC CRITERIA: Known allergy or hypersensitivity to AZD5305 or any of its excipients
* AZD5305 SPECIFIC CRITERIA: Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML
* AZD5305 SPECIFIC CRITERIA: Cardiovascular disease, QTc > 450 ms, or any factors that increase the risk of QTc prolongation or risk of arrhythmic events
* AZD5305 SPECIFIC CRITERIA: History of persisting (> 2 weeks) severe pancytopenia due to any cause (ANC < 0.5 x 10^9/L or platelets < 50 x 10^9/L)
* TREMELIMUMAB SPECIFIC CRITERIA: Medical co-morbidities that are deemed to make risk of surgery unacceptably high as determined by institutional standards
* TREMELIMUMAB SPECIFIC CRITERIA: Participants have received prior immunotherapy for the treatment of their PDAC
* TREMELIMUMAB SPECIFIC CRITERIA: Any unresolved toxicity Common Terminology Criteria for Adverse Events (CTCAE) > grade 2 from prior neoadjuvant therapy
* TREMELIMUMAB SPECIFIC CRITERIA: History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis, interstitial lung disease (ILD), pleural effusion, or pulmonary fibrosis diagnosed in the past 6 months prior to randomization
* TREMELIMUMAB SPECIFIC CRITERIA: Active or prior documented autoimmune or inflammatory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of all pharmacodynamic feasibility-evaluable participants within a study arm that have a measurable change in post-treatment tumor biology from baseline | Changes in tumor biology from baseline (i.e., Day 0) and on-treatment biopsy (i.e., 10 days from start of study intervention)
  Will be estimated with a 95% confidence interval (CI).

SECONDARY OUTCOMES:
Incidence of >= grade 3 toxicities for each assigned window treatment (as described in sub-protocol) | Up to 30 days
  Assessed per Common Terminology Criteria for Adverse Events version 5.0. The 95% CI will be reported with the point estimate of toxicity rate. All grade 3+ acute toxicities will also be summarized with its grade.

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Lopez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes